CLINICAL TRIAL: NCT01705548
Title: Phase I Dose Escalation Trial of Hypofractionated Radiosurgery for Large Brain Metastasis
Brief Title: Hypofractionated Stereotactic Radiosurgery in Treating Patients With Large Brain Metastasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bree Eaton, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00055063; NCI-2012-01933 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD2156-11 (Other: Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2012-10-10; First posted 2012-10-12 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Malignant Neoplasm to Brain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: Brain metastasis
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hypofractionated Radiosurgery (Experimental): HR (Hypofractionated Radiosurgery) delivered in 5 fractions, with a minimum of 2 and a maximum of 3 fractions being delivered per week, to patients with brain metastases or resection cavity greater than 3 cm and less than 6 cm.
  Dose escalation will proceed according to the Escalation with Overdose Control (EWOC) method with a planned total enrollment of 24 patients, in 8 patient cohorts with 3 patients per cohort. A 4 month observation period will occur for each completed cohort prior to dose escalation, with a goal timeline for trial completion of 4 years from first patient enrollment.
  Interventions: Radiation: Hypofractionated Radiosurgery

INTERVENTIONS:
Radiation: Hypofractionated Radiosurgery — Radiation Therapy will consist of partial brain irradiation delivered to the metastatic brain tumor or resection cavity, delivered in 5 treatments with 2-3 treatments delivered per week.

SUMMARY:
This phase I trial studies the side effects and best dose of hypofractionated radiosurgery in treating patients with large brain metastasis. Stereotactic radiosurgery can send x-rays directly to the tumor and cause less damage to normal tissue. Giving fractionated stereotactic radiosurgery may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To demonstrate the safety and feasibility of treating brain metastases or resection cavities greater than 3 cm with hypofractionated radiosurgery and to determine the maximum-tolerated radiation dose for hypofractionated radiosurgery (HR) delivered in 5 fractions, 2-3 fractions per week.

OUTLINE: This is a dose-escalation study.

Patients undergo hypofractionated stereotactic radiosurgery 2-3 times weekly (5 fractions total) for 2-3 weeks.

After completion of study treatment, patients are followed up at 1 month and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic proven diagnosis of solid tumor malignancy
* One brain metastasis or brain metastasis resection cavity with maximal diameter ≥ 3 cm (or ≥ 14 cc.) and ≤ 6 cm (or ≤ 113 cc.)
* Recursive partitioning analysis (RPA) class I-II/ Karnofsky Performance status (KPS) ≥ 70%

Exclusion Criteria:

* Prior stereotactic radiosurgery (SRS) to adjacent lesion such that planning target volume would have received more than 12 Gy
* RPA class III (KPS < 70%)
* Brain metastasis or resection cavity volume < 3 cm or > 6 cm
* Radiosensitive or non-solid (eg. small cell lung carcinomas, germ cell tumors, leukemias, or lymphomas) or unknown tumor histologies
* Concurrent chemotherapy (no chemotherapy starting 14 days before start of radiation)
* Evidence of leptomeningeal disease by magnetic resonance imaging (MRI) and/or cerebrospinal fluid (CSF) cytology
* Current pregnancy
* More than 8 weeks between resection and radiosurgical procedure
* Metastases to brain stem, midbrain, pons, or medulla or within 5 mm of the optic apparatus (optic nerves and chiasm)
* Inability to undergo MRI evaluation for treatment planning and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-09-24 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of hypofractionated radiosurgery defined as the highest dose level where a grade 3 or greater with an attribution score of ≥ 3 develops in ≤ 2 of 6 patients in a dose group | 4 months
  Graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. The rate of toxicities will be calculated with 95% confidence interval (CI).
Neurologic toxicity due to treatment, graded according to the CTCAE version 4.03 | Up to 2 years
  Calculated with 95% CI.

SECONDARY OUTCOMES:
Local control; lack of progression of disease in resection cavity as defined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria | 4 months
  The median time to local brain progression will be calculated by Kaplan-Meier method with 95% CI.
Distant control: lack of progression of disease in surrounding brain as defined by RECIST criteria | 4 months
  The median time to distant brain progression will be calculated by Kaplan-Meier method with 95% CI.
Freedom from failure/progression free survival | Up to 2 years
Overall survival (OS): death from any cause | Up to 2 years
  The median of OS time with 95% CI will be calculated by Kaplan-Meier method.
Long-term neurocognitive outcomes: using the Hopkins Verbal Learning Test-Revised (HVLT-R), Mini Mental Status Exam (MMSE) and Cognitive Functioning Subscale of the Medical Outcomes Scale (MOS) | Up to 2 years
  Neurocognitive effect will be regressed over time using generalized estimating equation (GEE) model. The population change over time (slope) will be estimated with 95% CI.
Quality of life (QOL) outcomes: using the quality of life questionnaire for the Functional Assessment of Cancer Therapy-Brain (FACT-Br). | Up to 2 years
  QOL outcomes will be regressed over time using GEE model. The population change over time (slope) will be estimated with 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Bree Eaton, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

DOCUMENTS (1):
  • Informed Consent Form (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT01705548/ICF_000.pdf